CLINICAL TRIAL: NCT01741441
Title: Study of Prognostic Factors for Long Term Results of Total Laparoscopic Fundoplication for Weakly Acidic or Mixed Reflux
Brief Title: Laparoscopic Total Fundoplication for Duodenogastroesophageal Reflux
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Fabrizio Rebecchi, Medical Doctor, University of Turin, Italy
Other Study IDs: LTF-2002-TO
Record Dates: First submitted 2012-11-25; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-11

CONDITIONS: Duodenogastric Reflux
Keywords: Duodenogastroesophageal reflux; Weakly acidic reflux; Gastric emptying; Laparoscopic fundoplication
MeSH Terms: conditions — Duodenogastric Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WAR and MR patients: Consecutive patients with MR and WAR selected for laparoscopic total fundoplication (LTF) were included in a prospective clinical study. Gastroesophageal function was assessed by clinical validated questionnaires, upper endoscopy, esophageal manometry and 24-h impedance pH monitoring before and 12 and 60 months after LTF. Gastric scintigraphy was preoperatively performed in all patients.
  Interventions: Procedure: laparoscopic total fundoplication

INTERVENTIONS:
Procedure: laparoscopic total fundoplication — LTF was performed using a standard five-trocar technique in all cases and carried out by two expert surgeons who had previously performed more than 50 laparoscopic fundoplications. A floppy 360° total fundoplication of 2-2,5 cm was constructed after full esophageal mobilization and posterior crural repair with nonabsorbable sutures.
  Other Names: Laparoscopic Nissen fundoplication; Laparoscopic 360° degree fundoplication

SUMMARY:
After laparoscopic total fundoplication (LTF) 12-15% of patients have persistent reflux symptoms and 20-25% develop gas-related symptoms. Reflux symptoms, gas bloating and inability to belch occurring after surgery have been associated with mixed (acid and weakly acid) (MR) or weakly acidic reflux (WAR). To date, few studies have evaluated functional outcome after LTF in patients with MR or WAR, with the majority reporting only short-term results.

It has been shown that delayed gastric emptying (DGE) might also be an important factor for abdominal distension and adverse outcome after LTF.9,10 However, the correlation between poor long-term outcome after LTF and DGE is controversial. In addition, the effect of DGE in patients with MR or WAR is poorly investigated.

DETAILED DESCRIPTION:
In the last years the study of gastro-oesophageal reflux has been revolutionized by the development of combined 24-h esophageal pH and multichannel intraluminal impedance (MII) monitoring.

Combined esophageal MII and pH-monitoring allow for the timed correlation of esophageal pH changes with reflux events and achieve high sensitivity for the detection of acid (pH <4), weakly acidic (pH 4-7) and weakly alkaline (pH >7) reflux episodes. Use of this technology is bringing into focus the potential role of weakly acidic and weakly alkaline reflux in symptoms that persist despite acid suppressive therapy or anti-reflux surgery.

ELIGIBILITY:
Inclusion Criteria:

- The study population consisted of consecutive patients with weakly acidic gastroesophageal reflux (GER) confirmed by 24 hour pH and impedance monitoring and eligible for laparoscopic antireflux surgery (LARS).

Exclusion Criteria:

- Exclusion criteria were presence of severe gastric emptying, functional heartburn, giant hiatal hernia, underlying primary esophageal motility disorder, American Association of Anaesthetists (ASA) score IV, previous upper abdominal surgery, and contraindications to pneumoperitoneum.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Between June 2002 and June 2007 188 patients with MR and WAR underwent LTF; 172 (91.5%) completed the 5-year protocol. Among them, forty-two (24.4%) had preoperative moderately delayed GE (DGE).
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2002-06; Primary Completion 2007-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
number of acidic and weakly acidic reflux | 60 months after LTF
  number of acidic and weakly acidic reflux at 24 hour pH impedance monitoring

SECONDARY OUTCOMES:
GERD Health related quality of Life score | 60 months after LTF
  Standard and previous validate questionnaire was employed in the study to assess gastroesophageal function and quality of life
Gastro-esophageal junction pressure | 60 months after surgery
  Gastroesophageal junction pressure was evaluated with esophageal manometry
Gastric emptying | 1 months before surgery
  Gastric emptying was evaluated with gastric scintigraphy before LTF

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Rebecchi, MD, Principal Investigator — University of Turin, Italy; Mario Morino, MD, Study Director — University of Turin, Italy; Marco Ettore Allaix, MD, Study Chair — University of Turin, Italy; Claudio Giaccone, MD, Study Chair — University of Turin, Italy
Locations (1):
- Digestive, Colorectal, Oncologic and Minimally Invasive Surgery, Department of Surgical Sciences, Turin, Italy

REFERENCES:
- [Background] Broeders JA, Mauritz FA, Ahmed Ali U, Draaisma WA, Ruurda JP, Gooszen HG, Smout AJ, Broeders IA, Hazebroek EJ. Systematic review and meta-analysis of laparoscopic Nissen (posterior total) versus Toupet (posterior partial) fundoplication for gastro-oesophageal reflux disease. Br J Surg. 2010 Sep;97(9):1318-30. doi: 10.1002/bjs.7174. PMID 20641062
- [Background] Broeders JA, Bredenoord AJ, Hazebroek EJ, Broeders IA, Gooszen HG, Smout AJ. Reflux and belching after 270 degree versus 360 degree laparoscopic posterior fundoplication. Ann Surg. 2012 Jan;255(1):59-65. doi: 10.1097/SLA.0b013e31823899f8. PMID 22167002
- [Background] Broeders JA, Bredenoord AJ, Hazebroek EJ, Broeders IA, Gooszen HG, Smout AJ. Effects of anti-reflux surgery on weakly acidic reflux and belching. Gut. 2011 Apr;60(4):435-41. doi: 10.1136/gut.2010.224824. Epub 2010 Dec 30. PMID 21193452
- [Background] Namasivayam V, Arora AS, Murray JA. Weakly acidic reflux. Dis Esophagus. 2011 Jan;24(1):56-62. doi: 10.1111/j.1442-2050.2010.01100.x. PMID 20659138
- [Background] Frazzoni M, Conigliaro R, Melotti G. Reflux parameters as modified by laparoscopic fundoplication in 40 patients with heartburn/regurgitation persisting despite PPI therapy: a study using impedance-pH monitoring. Dig Dis Sci. 2011 Apr;56(4):1099-106. doi: 10.1007/s10620-010-1381-4. Epub 2010 Aug 25. PMID 20737211
- [Background] Frazzoni M, Conigliaro R, Melotti G. Weakly acidic refluxes have a major role in the pathogenesis of proton pump inhibitor-resistant reflux oesophagitis. Aliment Pharmacol Ther. 2011 Mar;33(5):601-6. doi: 10.1111/j.1365-2036.2010.04550.x. Epub 2010 Dec 29. PMID 21198705
- [Background] Castell DO, Murray JA, Tutuian R, Orlando RC, Arnold R. Review article: the pathophysiology of gastro-oesophageal reflux disease - oesophageal manifestations. Aliment Pharmacol Ther. 2004 Dec;20 Suppl 9:14-25. doi: 10.1111/j.1365-2036.2004.02238.x. PMID 15527461
- [Background] Boeckxstaens GE. Review article: the pathophysiology of gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2007 Jul 15;26(2):149-60. doi: 10.1111/j.1365-2036.2007.03372.x. PMID 17593062
- [Background] Nakos A, Kouklakis G, Pitiakoudis M, Zezos P, Efraimidou E, Giatromanolaki A, Polychronidis A, Liratzopoulos N, Sivridis E, Simopoulos K. The histological and immunohistochemical aspects of bile reflux in patients with gastroesophageal reflux disease. Gastroenterol Res Pract. 2011;2011:905872. doi: 10.1155/2011/905872. Epub 2011 Jul 24. PMID 21822428
- [Background] Rebecchi F, Giaccone C, Farinella E, Campaci R, Morino M. Randomized controlled trial of laparoscopic Heller myotomy plus Dor fundoplication versus Nissen fundoplication for achalasia: long-term results. Ann Surg. 2008 Dec;248(6):1023-30. doi: 10.1097/SLA.0b013e318190a776. PMID 19092347
- [Background] Morino M, Giaccone C, Pellegrino L, Rebecchi F. Laparoscopic management of giant hiatal hernia: factors influencing long-term outcome. Surg Endosc. 2006 Jul;20(7):1011-6. doi: 10.1007/s00464-005-0550-6. Epub 2006 Jun 8. PMID 16763927
- [Derived] Rebecchi F, Allaix ME, Giaccone C, Morino M. Gastric emptying as a prognostic factor for long-term results of total laparoscopic fundoplication for weakly acidic or mixed reflux. Ann Surg. 2013 Nov;258(5):831-6; discussion 836-7. doi: 10.1097/SLA.0b013e3182a6882a. PMID 24045453